CLINICAL TRIAL: NCT03483896
Title: Pilot Study to Examine the Effects of Indoor Daylight Exposure on Depression and Other Neuropsychiatric Symptoms in People Living With Dementia in Long Term Care Facilities
Brief Title: Pilot Study to Examine Health Effects of Daylight Exposure on Dementia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Kyle Konis, Assistant Professor, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UP-16-00487
Record Dates: First submitted 2018-03-21; First posted 2018-03-30 (Actual); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2018-12

CONDITIONS: Dementia; Depression; Behavior Disorders
MeSH Terms: conditions — Dementia; Depression; Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): At the 4 facilities in the control arm, participants received the usual care. During the period from 8:00 - 10:00 AM each day, the control group was taken to a similar sized area indoors (without daylight) for socialization under typical electrical lighting conditions.
- Daylight Intervention (Active Comparator): At the 4 facilities in the active light intervention arm, staff increased the daylight exposure of participants by taking them to the perimeter zone of a daylit room from 8:00 to 10:00 AM for socialization over a period of 12 weeks. The perimeter zone was defined to be the region of the room within 3 meters from windows. The intervention was administered each day (7 days / week) over the duration of the study.
  Interventions: Other: Daylight Intervention

INTERVENTIONS:
Other: Daylight Intervention — Staff increased the daylight exposure of participants by taking them to the perimeter zone of a daylit room from 8:00 to 10:00 AM for socialization over a period of 12 weeks. The perimeter zone was defined to be the region of the room within 3 meters from windows. The intervention was administered each day (7 days / week) over the duration of the study.
  Arms: Daylight Intervention

SUMMARY:
This study is designed to test the hypothesis that an intervention increasing exposure to daylight indoors will reduce depression and other neuropsychiatric symptoms among people living with dementia in long term care facilities.

DETAILED DESCRIPTION:
Exposure to sufficient daylight indoors is a novel and potentially effective nonpharmacological treatment option for reducing depression and other neuropsychiatric symptoms for people living with dementia in long term care facilities. However, there are currently no minimum requirements for daylight access in care facilities. In urban settings, it is common for residents to spend the majority of the day indoors, illuminated by electrical light sources that deliver light with significantly lower intensities and reduced spectrum compared with daylight.

A 12-week pilot study was conducted in 8 dementia care facilities involving (n = 83) participants addressing the hypothesis that an intervention increasing indoor exposure to daylight will reduce depression and other neuropsychiatric symptoms. At 4 facilities, staff was enlisted to increase daylight exposure by taking participants to a perimeter room with daylight exposure for socialization in the morning (8:00 - 10:00 AM) each day. At the other 4 facilities, a control group were taken to a similar sized area without daylight for socialization under typical electrical lighting conditions. Outcome measures for depression and other neuropsychiatric symptoms were taken at the beginning and end of the 12-week study.

ELIGIBILITY:
Inclusion Criteria:

* Residents were recruited according to the trial inclusion criteria: 1) Alzheimer's disease and related dementias (ADRD) diagnosis, 2) no physical co-morbidities that precluded participation in the daily group intervention, and 3) a Mini-Mental State Exam (MMSE) score of 10 or higher

Exclusion Criteria:

* physical co-morbidities that precluded participation in the daily group intervention

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Konis, Ph.D, Principal Investigator — University of Southern California
Locations (8):
- United States (8):
  - Alhambra Dementia Care, Alhambra, California
  - Sierra Vista Memory Care Community, Azusa, California
  - Calabasas Memory Care Community, Calabasas, California
  - Costa Mesa Dementia Care, Costa Mesa, California
  - Los Angeles Dementia Care (Beverly Place), Los Angeles, California
  - Redondo Beach Dementia Care (Beach Cities), Redondo Beach, California
  - San Juan Capistrano Memory Care Community, San Juan Capistrano, California
  - Tustin Hacienda Memory Care Community, Tustin, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Daylight Intervention
Started | 33 | 50
Completed | 31 | 46
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Daylight Intervention | Total
Number analyzed (Participants) | 31 | 46 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 84.7 (7.3) | 85.6 (6.9) | 85.3 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 31 | 56
  Male | 6 | 15 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White race | 29 | 42 | 71
  Ethnicity: Non-white race | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 31 | 46 | 77
Cornell Scale for Depression in Dementia (CSDD) [Mean (Standard Deviation); unit: units on CSDD scale] — The Cornell Scale for Depression in Dementia (CSDD) was used to measure depression. The CSDD is designed for the assessment of depression in older people with dementia who can at least communicate basic needs. The CSDD scale ranges from 0 to 38, with higher scores indicating higher levels of depression. Scores above 10 indicate a probable major depression. Scores above 18 indicate a definite major depression. Scores below 6 are associated with absence of significant depressive symptoms. Population: Included patients with CSDD obtained within 4 months of start of study, leading to 28 analyzed for the control group (of 31) and 38 analyzed for the Daylight Intervention group (of 46). Baseline means and SDs reported here do not account for clustering within facility.
  units on CSDD scale
    number analyzed (Participants) | 28 | 38 | 66
    (all) | 4.4 (4.5) | 5.0 (5.4) | 4.4 (4.5)
Neuropsychiatric Inventory Nursing Home Version (NPI-NH) [Mean (Standard Deviation); unit: units on NPH-NH scale] — The NPI-NH includes ten behavioral areas and two types of neurovegetative changes. Each of the 12 areas is scored on a subscale ranging from 0-12, where higher scores indicate greater neuropsychiatric symptomatology. A summary score is obtained from summing all 12 subscale scores. The summary score ranges from 0 - 144, where higher scores indicate greater neuropsychiatric symptomatology.
  Baseline means and SDs reported here do not account for clustering within facility.
  units on NPH-NH scale | 16.3 (14.5) | 16.0 (19.1) | 16.1 (17.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cornell Scale for Depression in Dementia (CSDD)
Description: The Cornell Scale for Depression in Dementia (CSDD) was used to measure depression. The CSDD is designed for the assessment of depression in older people with dementia who can at least communicate basic needs. The CSDD scale ranges from 0 to 38, with higher scores indicating higher levels of depression. Scores above 10 indicate a probable major depression. Scores above 18 indicate a definite major depression. Scores below 6 are associated with absence of significant depressive symptoms.
Time Frame: A CSDD score was taken at the beginning of the 12-week study and once again at the end of the 12-week study.
Population: Included patients with CSDD obtained within 4 months of start of study, leading to 28 analyzed for the control group (of 31) and 38 analyzed for the Daylight Intervention group (of 46). Baseline means and SDs reported here do not account for clustering within facility.
Measure: Mean (Standard Error); unit: units on CSDD scale
Arm/Group | Control | Daylight Intervention
Number analyzed (Participants) | 28 | 36
units on CSDD scale | 1.5 (1.0) | -2.0 (0.9)
Statistical Analysis 1: Comparison: Control vs Daylight Intervention; Test type: Superiority; p = 0.01, Mixed Models Analysis; Mean Difference (Final Values) = -3.5

2. Secondary Outcome: Change in Neuropsychiatric Inventory Nursing Home Version (NPI-NH)
Description: The Neuropsychiatric Inventory Nursing Home Version (NPI-NH) was used to measure neuropsychiatric symptomatology. The NPI-NH is a scale designed for assessment of people with dementia residing in extended care facilities. The NPI-NH includes ten behavioral areas (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior) and two types of neurovegetative changes (sleep and nighttime behavior disorders, appetite and eating disorders). Each of the 12 areas is scored on a subscale ranging from 0-12, where higher scores indicate greater neuropsychiatric symptomatology. A summary score is obtained from summing all 12 subscale scores. The summary score ranges from 0 - 144, where higher scores indicate greater neuropsychiatric symptomatology.
Time Frame: A NPI-NH score was taken at the beginning of the 12-week study and once again at the end of the 12-week study.
Measure: Mean (Standard Error); unit: Units on NPH-NH scale
Arm/Group | Control | Daylight Intervention
Number analyzed (Participants) | 31 | 46
Units on NPH-NH scale | 3.1 (3.2) | -2.8 (2.9)
Statistical Analysis 1: Comparison: Control vs Daylight Intervention; Test type: Superiority; p = 0.17, Mixed Models Analysis; Mean Difference (Final Values) = -6.0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Control | Daylight Intervention
All-Cause Mortality (participants affected / at risk) | 2/33 | 1/50
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/50
Other Adverse Events (participants affected / at risk) | 0/33 | 0/50

LIMITATIONS AND CAVEATS:
Scheduling problems with baseline measures led to CSDD scores from health records being used for some participants with scoring dates that predated the start of the study by up to 4 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03483896/Prot_SAP_000.pdf